CLINICAL TRIAL: NCT05433298
Title: Multicenter Phase I/IIa Study of Mesenchymal Stromal Cells for the Treatment of Patients With SARS-CoV-2 Pneumonia.
Brief Title: Mesenchymal Stromal Cells for the Treatment of Patients With COVID-19.
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No patient could be included because there was a decrease in the number of patients with complications due to COVID-19. Also, a Brazilian government agency approved this clinical trial, and the project execution period ended in March 2023.
Sponsor: Paulo Brofman (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor-Investigator, Paulo Brofman, Principal Investigator, Pontifícia Universidade Católica do Paraná
Organization: Pontifícia Universidade Católica do Paraná (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MSC SARS-CoV-2; U1111-1267-1200 (Other: UTN - WHO International Clinical Trials Registry Platform); 31935420.7.1001.0020 (Other: CAAE - Certificado de Apresentação para Apreciação Ética)
Record Dates: First submitted 2022-05-19; First posted 2022-06-27 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: COVID-19 Pneumonia; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Patient: Intravenous infusion of single-dose of Mesenchymal stem cells (MSCs)
  Interventions: Biological: Mesenchymal stem cell
- Placebo (Placebo Comparator): Intravenous infusion of single-dose of Ringer's lactate, albumin and heparin solution
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Mesenchymal stem cell — Administration of advanced cell product
  Arms: Treatment
Other: Placebo — Ringer's lactate, albumin and heparin solution
  Arms: Placebo

SUMMARY:
The purpose of this study is evaluate the feasibility, safety and potential efficacy of an advanced cell therapy product for the treatment of patients with SARS-CoV-2 pneumonia.

DETAILED DESCRIPTION:
Forty patients with COVID-19 will receive an intravenous infusion of one dose of 1.000.000 umbilical cord mesenchymal cells per kilo of the patient. Twenty patients will receive a placebo (Ringer's lactate solution, albumin and heparin). Conventional treatment will be performed together with the infusion of cells, during the study period. The evaluation times will be at pre-infusion, 6 and 24 hours, days 5 and 28, 3 and 6 months. The patient exams performed: serology, biochemistry, blood count and blood gas analysis, metabolomics/proteomics, antibody evaluation, electrocardiogram, CT-scan and X-ray, cytokines, viral load, cytometry, and clinical evaluation. The patients will be evaluated all the time, during hospitalization period, to assess adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes;
* aged 18 to 79 years old;
* hospitalized patients;
* radiological diagnosis of viral pneumonia;
* virological diagnosis of SARS-CoV-2 infection;
* with noninvasive ventilatory support;
* C-reactive protein and ferritin above the reference value considered normal;
* assent confirmed to participate in the study.

Exclusion Criteria:

* Contraindications for use of corticosteroids;
* immunosuppressive, cytotoxic and antiviral treatment, experimental medications and chronic corticosteroid use;
* morbid obesity (BMI> 35);
* multiple organ dysfunction syndrome;
* pre-malignant neoplastic conditions with life expectancy lower than 1 year old;
* pre-existing chronic illnesses like chronic dialysis kidney disease, chronic liver disease, congestive heart failure Class IV; pulmonary hypertension (WHO Class III/IV);
* pre-existing or current thromboembolic pathology;
* transplanted patients;
* pre-existing severe allergic reaction;
* history of HIV and tuberculosis;
* enrollment in another clinical trial;
* pregnancy or breastfeeding.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-11-26 (Estimated); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Safety of intravenously infused UCT-MSC suspension | After first cell infusion until the end of study. The clinical follow-up of patients will be one year after the transplant.
  The primary expected outcome is the safety and tolerability of using intravenously infused UTC-MSC suspension in patients with pneumonia caused by SARS-CoV-2. This outcome will be evaluated by recording adverse events that must be reported throughout the study period.

SECONDARY OUTCOMES:
Pulmonary function test to evaluate the improvement of respiratory function | Pre-infusion, on days 5 and 28, 3 and 6 months.
  Evaluation of lung function.
Radiography to evaluate the improvement of respiratory function | Pre-infusion, on days 5 and 28, 3 and 6 months.
  Evaluation of pulmonary function using breathing chest radiography. Assessment of peripheral opacities, interstitial and airspace opacities, diffuse airspace opacities, interstitial opacities, lobar consolidation, atelectasis, cavities, pulmonary cysts, and emphysema.
6-minute walk to evaluate the improvement of respiratory function | Pre-infusion, on days 5 and 28, 3 and 6 months.
  Distance covered by the patient in a period of 6 minutes.
Decrease on days of non-invasive mechanical ventilation | Six hours after infusion, days 1, 5 and 28, 3 and 6 months.
  Analysis of ventilatory parameters and arterial blood gas analysis.
Biochemical tests to evaluate the improvement of laboratory parameters | Pre-infusion, on days 1, 5 and 28, 3 and 6 months.
  D-dimer, C-reactive protein, erythrocyte sedimentation rate, ferritin, creatine, urea, saline, potassium, bilirubin, total protein and fractions, albumin, globulin, oxalacetic transaminase, pyruvic transaminase, lactate dehydrogenase, creatine phosphokinase, troponin I, coagulogram.
Blood count to evaluate the improvement of laboratory parameters | Pre-infusion, on days 1, 5 and 28, 3 and 6 months.
  Red blood cells, hemoglobin, hematocrit, total leukocytes, basophil, eosinophil, neutrophil, lymphocytes, monocytes, platelets.
Viral load to evaluate the improvement of laboratory parameters | Pre-infusion, on days 1, 5 and 28, 3 and 6 months.
  Expression of the RpRd gene.
Cytokine dosage to evaluate inflammatory parameters | Pre-infusion, on days 1, 5 and 28, 3 and 6 months.
  Granulocyte-macrophage colony-stimulating factor (GM-CSF), interleukin (IL) -2, IL-6, IL-7, IL-8, tumor necrosis factor (TNF) α, monocyte chemoattractant protein-1 (MCP1/CCL2) and macrophage inflammatory protein 1-alpha (MIP1a/CCL3).
Decrease in hospital stay | From admission to discharge, or a maximum of 6 months.
  Evaluation of hospitalization days.
Computed tomography score to evaluate the improvement of pulmonary function | Pre-infusion, on days 5 and 28, 3 and 6 months.
  Chest computed tomography evaluation will analyze the following characteristics: ground glass opacities, linear opacities, consolidation, interlobular septal thickening, crazy-paving pattern, subpleural lines, bronchial wall thickening, lymph node enlargement and pleural effusion. Lesions will quantify by assigning a score to all abnormal areas involved. Each lobe will assigned a score of 0 (0% involvement), 1 (1-25% involvement), 2 (26-50% involvement), 3 (51-75% involvement) or 4 (76%-100% involvement). The total score will be the sum of all lobes, ranging from 0 to 25.
Reduction in the percentage of intubated patients | After first cell infusion until six months after the transplant.
  Clinical evaluation of patients.
Decrease in mortality | After first cell infusion until the end of study. The clinical follow-up of patients will be six months after the transplant.
  Evaluation of the number of patients who died during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo R Brofman, phD, Principal Investigator — Pontifícia Universidade Católica do Paraná
Locations (1):
- Paulo Roberto Slud Brofman, Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rebelatto CLK, Senegaglia AC, Franck CL, Daga DR, Shigunov P, Stimamiglio MA, Marsaro DB, Schaidt B, Micosky A, de Azambuja AP, Leitao CA, Petterle RR, Jamur VR, Vaz IM, Mallmann AP, Carraro Junior H, Ditzel E, Brofman PRS, Correa A. Safety and long-term improvement of mesenchymal stromal cell infusion in critically COVID-19 patients: a randomized clinical trial. Stem Cell Res Ther. 2022 Mar 21;13(1):122. doi: 10.1186/s13287-022-02796-1. PMID 35313959
- [Background] Senegaglia AC, Rebelatto CLK, Franck CL, Lima JS, Boldrini-Leite LM, Daga DR, Leitao CA, Shigunov P, de Azambuja AP, Bana E, Marsaro DB, Schaidt B, Micosky A, Jamur VR, Schluga Y, Vaz IM, Ribeiro LL, Correa A, Brofman EPRS. Combined Use of Tocilizumab and Mesenchymal Stromal Cells in the Treatment of Severe Covid-19: Case Report. Cell Transplant. 2021 Jan-Dec;30:9636897211021008. doi: 10.1177/09636897211021008. PMID 34074163
- See also: UC-MSCs infusion is safe and can play an important role as an adjunctive therapy, both in the early stages, preventing severe complications and in the chronic phase with postacute sequelae reduction in critically ill COVID-19 patients. — https://pubmed.ncbi.nlm.nih.gov/35313959/
- See also: The combination of tocilizumab and UC-MSC proved to be safe, with no adverse effects, and the results of this case report prove to be a promising alternative in the treatment of patients with severe acute respiratory syndrome due to SARS-CoV-2. — https://pubmed.ncbi.nlm.nih.gov/34074163/